CLINICAL TRIAL: NCT06700057
Title: Optimisation and Safety of an Innovative Nuclear Medicine Treatment: Clinical and Dosimetric Study of Patients Treated With 177Lu-PSMA-617 for Prostate Cancer.
Brief Title: Clinical and Dosimetric Study of Patients Treated With 177Lu-PSMA-617 for Prostate Cancer.
Acronym: DOSIPROSTATE
Status: Recruiting | Type: Observational
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Other Study IDs: IB 2024 - DOSIPROSTATE
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer; Metastasis
Keywords: Radiopharmaceutical drug
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Single-centre, retrospective and prospective observational study. This study aims to evaluate the dose delivered by radiation to the tumour and organs at risk, as a factor predicting response and the appearance of toxicities. Dosimetric calculations are made for each treatment using scintigraphic images acquired following injection of 177Lu-PSMA-617.

DETAILED DESCRIPTION:
The management of patients and the administration of treatment with 177Lu-PSMA are carried out in the usual way in the nuclear medicine department of the Institut Bergonié, and are not modified in any way.

The treatment regimen is standard, with 6 cycles spaced 6 weeks apart at a fixed dose of 7.4 GBq. Patients are selected on the basis of a 68Ga-PSMA-11 PET/CT scan to assess whether PSMA is properly expressed.

Only data are collected for the study and they are derived from the usual management of patients treated with 177Lu-PSMA at the Institut Bergonié: information on the treatment, anatomical data and 177Lu-PSMA fixation in lesions and tissues, scintigraphic images acquired post-treatment, data on monitoring the effects of the treatment, 68Ga-PSMA PET/CT images.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 18 and over.
2. Patient with indication for or having started or completed treatment with 177Lu-PSMA-617 since 01/11/2023:

   1. Progressive, metastatic, castration-resistant prostate cancer,
   2. overexpressing prostate specific membrane antigen (PSMA)
   3. treated with taxane chemotherapy and at least one 2nd generation hormone therapy (apalutamide, enzalutamide, darolutamide, abiraterone-prednisone).
3. Patient able to lie still for 1 hour for image acquisition.
4. Patient's place of residence < 2 hours' drive from the Institut Bergonié.
5. Patient has not expressed any opposition to the use of his/her medical data for research purposes.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic castration-resistant prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Median of total absorbed-dose of 177Lu-PSMA-617 at total tumor volume as a function of prostate-antigen specific (PSA) response | From pre-treatment baseline to the end of treatment and after the end of treatment, i.e approximately 10 months.
  To assess the association between the total absorbed-dose of treatment at total tumor volume and the efficacy of treatment in terms of PSA response rate (PSA50-RR).
  PSA50-RR is defined by the proportion of patients with a decrease ≥ 50% in PSA concentration from pre-treatment baseline, confirmed by a subsequent PSA assessment performed at least 3 weeks later.
  Absorbed-dose of treatment at total tumor volume, expressed in Gray (Gy), is calculated for each course of 177Lu-PSMA-617 (every 6 weeks +/- 1 week) from SPECT/CT images acquired post administration with PlanetDose software (DOSIsoft). The total absorbed dose in Gray (Gy) is defined by the sum of absorbed doses over all courses of treatment performed.

SECONDARY OUTCOMES:
Median of total absorbed-dose of 177Lu-PSMA-617 at total tumor volume as a function of best overall response (RECIST v1.1) | From pre-treatment baseline to the end of treatment and after the end of treatment, i.e approximately 10 months.
  To assess the association between the total absorbed-dose of treatment at total tumor volume and the efficacy of treatment in terms of best overall response according to RECIST v1.1. Best overall response is defined as the best response evaluated according to RECIST v1.1, observed between initiation and end of treatment. It is determined once all data for the same patient are known. Absorbed-dose of treatment at total tumor volume, expressed in Gray (Gy), is calculated for each course of 177Lu-PSMA-617 (every 6 weeks +/- 1 week) from SPECT/CT images acquired post administration with PlanetDose software (DOSIsoft). The total absorbed dose in Gray (Gy) is defined by the sum of absorbed doses over all courses of treatment performed.
Median of total absorbed-dose of 177Lu-PSMA-617 at total tumor volume as a function of objective functional response (nuclear physician assessment))) | From pre-treatment baseline to the end of treatment (Dose) and at the end of treatment (bjective functional response), i.e approximately 10 months.
  To assess the association between the total absorbed-dose of treatment at total tumor volume and the efficacy of treatment in terms of objective functional response on 68Ga-PSMA-11 PET, defined as complete response or partial response, based on image interpretation by the nuclear physician. Absorbed-dose of treatment at total tumor volume, expressed in Gray (Gy), is calculated for each course of 177Lu-PSMA-617 (every 6 weeks +/- 1 week) from SPECT/CT images acquired post administration with PlanetDose software (DOSIsoft). The total absorbed dose in Gray (Gy) is defined by the sum of absorbed doses over all courses of treatment performed.

CONTACTS AND LOCATIONS:
Overall Officials: Nadège ANIZAN, Study Director — Institut Bergonié
Locations (1):
- Institut Bergonie, Bordeaux, France